CLINICAL TRIAL: NCT02191059
Title: Single Arm, Phase II Clinical Study of Intermittent High Dose of Icotinib in Combination With Docetaxel as Second-line Treatment for Non-small Cell Lung Cancer Patients With Wild Type EGFR:
Brief Title: Phase II Clinical Study of Intermittent High Dose of Icotinib in Combination With Docetaxel to Treat Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Zhehai Wang, Vice President, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Icotinib
Record Dates: First submitted 2014-07-13; First posted 2014-07-15 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non Small Cell Lung Cancer; Wild Type EGFR; Icotinib; Second-line Treatment
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — icotinib; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intermittent High Dose of Icotinib (Experimental): Intermittent High Dose of Icotinib in Combination With Docetaxel:
  Icotinib 625mg tablet b ymouth three times per day for day1-2, Docetaxel 75mg/m2 injection intravenous drip for day 3, 3 weeks as 1 cycle
  Interventions: Drug: Icotinib; Drug: Docetaxel

INTERVENTIONS:
Drug: Icotinib
Drug: Docetaxel
  Other Names: Taxotere, Docecad

SUMMARY:
1. There is as yet no optimal treatment regimen for patients with epidermal growth factor receptor (EGFR) gene wild type non-small-cell lung cancer (NSCLC) .
2. Icotinib is a new type of small molecule EGFR TKI, developed and patented by Zhejiang BetaPharma Co., Ltd.(Hangzhou, Zhejiang, China, Patent No. WO2003082830). It has the similar anti-tumor activity with gefitinib, erlotinib. Pre-clinical studies showed icotinib could significantly inhibit the EGFR tyrosine kinase activity. Notably, anti-tumor activities were observed in patients with advanced NSCLC.
3. In this study, we will evaluate the efficiency of intermittent high dose of Icotinib in combination with Docetaxel as second-line treatment for NSCLC patients with wild type EGFR. The overall response rate(ORR),progression free survival(PFS) ,overall survival(OS) and health related quality of life(HRQoL) will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed stage IIIB/IV NSCLC patients progressing after first-line chemotherapy;
* Patients must have stopped prior platinum-based therapy at least four weeks prior to enroll and fully recovered from chemotherapy-induced toxicity;
* Age: 18-70 years old;
* Patients with wild-type EGFR;
* With a histologically or cytologically confirmed measurable disease (longest diameters >=10mm with Spiral computed tomography (CT)and >=20mm with conventional CT) according to Response Evaluation Criteria in Solid Tumors (RECIST Criteria);
* Patients must have Eastern Cooperative Oncology Group(ECOG)Performance Status of 0-2;
* Must have an expected survival time of at least 12 weeks;
* Patients should have adequate bone marrow function defined as an absolute peripheral neutrophil count (ANC) of ≥1.5 ´ 109/L, platelet count of ≥ 75´ 109/L; Hemoglobin(Hb) ≥ 9g/dL;
* adequate hepatic function: bilirubin ≤2x the upper limit of normal, glutamic-oxaloacetic transaminase(AST )and glutamate pyruvate transaminase(ALT)≤2x the upper limit of normal (≤5x the upper limit of normal if evidence of liver metastases);
* adequate renal function: bilirubin serum creatinine ≤1.5 x the upper limit of normal;
* No malabsorption or other gastrointestinal disorders affecting drug absorption;
* Female patients of childbearing potential must have a negative serum or urine pregnancy test within 7 days prior to study entry.Male patients must use at least one reliable form of contraception during treatment and within 3 months after treatment;
* Patients have provided a signed Informed Consent Form.

Exclusion Criteria:

* Experience of Anti-EGFR Monoclonal Antibody or small molecular compounds therapy such as gefitinib, cetuximab, erlotinib or trastuzumab;
* Concomitant use with phenytoin, carbamazepine, rifampicin, phenobarbital or St. John's Wort;
* Allergic to icotinib or any of the excipients of this product.
* Prior chemotherapy with any paclitaxel agents;
* Central nervous system (CNS) metastases without radiotherapy and/or surgery;
* Evidence of clinically active Interstitial lung diseases;
* Severe systemic disease out of control such as unstable or uncompensated respiratory,cardiac,liver,renal diseases;
* Patient has a concurrent malignancy or has a malignancy within 5 years of study enrollment, (with the exception of non melanoma skin cancer or cervical carcinoma in situ);
* Psychiatric illness that would prevent the patient from giving informed consent;
* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the subject to participate in the study;
* Patient is concurrently using other approved or investigational antineoplastic agent;
* Pregnant or lactating women;
* Positive epidermal growth factor receptor mutation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate(ORR) | 10-12 months

SECONDARY OUTCOMES:
Progression Free Survival(PFS) | 10-12 months
Overall Survival(OS) | 10-12momths
Health Related Quality of Life(HRQoL) | 10-12months

CONTACTS AND LOCATIONS:
Overall Officials: Zhehai Wang, MD, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Shandong Cancer Hospital and Institute, Jinan, Shandong, China